CLINICAL TRIAL: NCT06845111
Title: The Effect of Therapeutic Play-Based Intervention Programme (TOTEM) Applied to 4-6 Age Group Earthquake Victims Living in Kahramanmaraş on Children's Psychosocial Well-Being
Brief Title: Therapeutic Play and Its Effect on Children's Psychosocial Well-Being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Collaborators: Kahramanmaraş İstiklal University (Other)
Responsible Party: Principal Investigator, Sinem Yalnızoglu Caka, Assoc. Prof., Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023/15/15; 123S913 (Other Grant/Funding Number: TÜBİTAK)
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2024-05

CONDITIONS: Therapeutic Play; Psychosocial Well-being; Nursing Care
Keywords: Child; anxiety; psychosocial status; disturbance; nursing care
MeSH Terms: conditions — Anxiety Disorders | interventions — Play Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single (third party blinding- Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Group receiving Therapeutic Play (Experimental): The Therapeutic Play-Based Intervention Programme (TOTEM) designed for the research was carried out with the children in the intervention group on the determined days and hours. The children were administered the post-test immediately after the end of the programme and then the retention test at the end of the first month.
  Interventions: Other: Therapeutic play
- Control Group (No Intervention): Control group (routine education programme): The children in the control group were administered a pre-test in the kindergartens they were currently attending (which were included in daily routine life, games, etc. by preschool teachers living in the city), a post-test after five weeks in parallel with the study group, and then a retention test at the end of the first month. Considering ethical principles, the TOTEM programme was also applied to the children in this group after the study was completed.

INTERVENTIONS:
Other: Therapeutic play — In this context, the pre-school teachers in the container area were contacted and the sessions were held every Wednesday-Thursday (8 sessions in total) for 5 weeks, taking into account their availability hours. Children were included in the programme in groups of 12. Before data collection, the necessary materials were provided and stored in an empty container. It was found appropriate to complete the trainings in kindergartens located in the container city (4). A total of 3 evaluations were carried out: a post-test immediately after the end of the programme and a retention test at the end of the first month.
  Arms: Experimental: Group receiving Therapeutic Play

SUMMARY:
The aim of this study was to evaluate the effectiveness of the Therapeutic Play-Based Intervention Programme (TOTEM), which was developed to reduce the negative psychosocial effects of the earthquake in children aged 4-6 years, and its effect on children's psychosocial well-being.

DETAILED DESCRIPTION:
Earthquakes are among the most impressive geological processes and are defined as an unpredictable natural disaster due to their destructive effects on people and structures. In Turkey, a 7.7-magnitude earthquake occurred on 6 February 2023 at 04.17 local time, centred in Kahramanmaraş, and another 7.6-magnitude earthquake occurred about nine hours later. In addition, more than 1000 aftershocks were recorded in the region and these events further increased the scale of the disaster. Earthquakes have the potential to have profound and traumatic effects on people's psychological functioning. Children are particularly affected by these effects due to their vulnerability during natural disasters. Children who experience disasters may face various problems in physical, cognitive and socio-emotional development.

Therapeutic play intervention is based on the belief that play is a universal language that allows children to easily express their feelings and thoughts. This approach is an effective strategy that helps the child to explore their problems, seek solutions, express their feelings and emotional regulation. It also promotes cognitive development, reduces anxiety and stress, and increases confidence.

Providing appropriate support to children after a traumatic event such as an earthquake is critical for preventing future psychological problems. In this context, providing children with supportive approaches such as play therapy and conducting these methods by expert teams can contribute to children's well-being. Therapeutic games play an important role by providing a universal language for children to express their emotions and cope with stress.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 4-6
* Having literate parents
* Having adequate Turkish receptive-expressive language skills
* Not having a previously diagnosed psychiatric problem declared by the parents
* Not having participated in a training programme on psychosocial well-being before
* Not attending any pre-school education institution at the time of the training
* Volunteering to participate in the study by themselves and their parents

Exclusion Criteria:

* The participant wants to leave the study
* The participant has not participated in one or more of the trainings to be given within the scope of the programme
* The participant shows any diagnosed atypical development
* Children who show a level of resistance that disrupts their adaptation to normal life in pre-tests, during the study or in post-tests, children with anxiety disorder or other psychiatric problems

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Anxiety Scale in Preschool Children | A total of 3 evaluations will be made: before the programme starts, the post-test immediately after the end of the programme and the retention test at the end of the first month.
  The Anxiety Scale in Preschool Children (Spence et al., 2001) developed by Spence, Rapee, McDonald, Ingram (2001) was adapted into Turkish by Şahin (2020). While the original scale had 28 items measuring social anxiety, separation anxiety, fear of physical injury, general anxiety and obsessive-compulsive disorder, Şahin added 5 items related to post-traumatic stress disorder while adapting it to Turkish and validity and reliability studies were conducted with these items. The scale is a 5-point scale and each item is scored between 0 and 4. A total score can be obtained from the scale. A high score on the scale indicates that anxiety in preschool children is high, while a low score indicates that anxiety in preschool children is low. Within the scope of the reliability of the scale, Cronbach's Alpha coefficient was calculated as 0.93 (Şahin, 2020). For this study, Cronbach's Alpha coefficient was calculated as 0.91.
Psychosocial Status Assessment Scale for 3-6 Year Old Children (Parent Form) | A total of 3 evaluations will be made: before the programme starts, the post-test immediately after the end of the programme and the retention test at the end of the first month.
  Psychosocial Situation Rating Scale (PSRS) was developed by Güneş-Şan and Altay and is a measurement tool consisting of 31 items that measures Psychosocial Situation Rating based on parental report in children aged 3-6 years. For each item in the PSDD, there are 5-point Likert type options 0-'never', 1-'rarely', 2-'sometimes', 3-"often", 4-'always'. Based on the score given for each item, a minimum score of '0' and a maximum score of '124' can be obtained from the questionnaire. A low total score indicates that there is no risk for psychosocial problems in the child, while a high score indicates that there is a risk for psychosocial problems. Within the scope of the reliability of the scale, Cronbach's Alpha coefficient was calculated as 0.83 and test-retest reliability was calculated as 0.957 (Güneş-Şan & Altay, 2021). For this study, Cronbach's Alpha coefficient was calculated as 0.88.
Sleep Disturbance Scale for Children | A total of 3 evaluations will be made: before the programme starts, the post-test immediately after the end of the programme and the retention test at the end of the first month.
  The scale developed by Bruni et al. (1996) was adapted into Turkish and the validity and reliability study was conducted by Ağça-Bilmenoğlu (2019). The scale developed to investigate sleep disorders in children consists of 26 items and each question is scored between 1-5. The measurement tool includes questions measuring sleep initiation and maintenance problems, sleep breathing disorders, sleep-wake disorders, sleep-wake transition disorders, excessive sleepiness disorders and excessive sweating during sleep. The scores that can be obtained from the scale vary between 26 and 130, and high scores are interpreted as a high degree of sleep disorder. Within the scope of the reliability of the scale, Cronbach's Alpha coefficient was calculated as 0.84 and test-retest reliability as 0.79 (Ağça-Bilmenoğlu, 2019). For this study, Cronbach's Alpha coefficient was calculated as 0.85.

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University, Kocaeli, Izmit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park EJ, Lee MS, Bae SM, Kim HS, Hong M, Kim E, Lee SK, Kim J, Bhang SY. Promising Effect of the Children in Disaster: Evaluation and Recovery Intervention on Trauma Symptoms and Quality of Life for Children and Adolescents: A Controlled Study. Psychiatry Investig. 2024 Feb;21(2):123-132. doi: 10.30773/pi.2023.0202. Epub 2024 Feb 8. PMID 38321890
- [Background] Wong CL, Ip WY, Kwok BMC, Choi KC, Ng BKW, Chan CWH. Effects of therapeutic play on children undergoing cast-removal procedures: a randomised controlled trial. BMJ Open. 2018 Jul 5;8(7):e021071. doi: 10.1136/bmjopen-2017-021071. PMID 29980545
- [Background] Juwita, H. 2019. "Effectiveness of multimodal interventions play therapy: Colouring and origami against anxiety levels in toddler ages," Journal of Health Science and Prevention, 3(3S), 46-51.
- [Background] Silva, L., Oliveira, C., Oliveira, J., Bandeira, P., Matos, J., Gomes, E., et al. 2022. "Use of therapeutic play in nursing care for school-age children: a scoping review," Preprints (2022).
- [Background] Satapathy S, Dang S, Sagar R, Dwivedi SN. Resilience in Children and Adolescents Survived Psychologically Traumatic Life Events: A Critical Review of Application of Resilience Assessment Tools for Clinical Referral and Intervention. Trauma Violence Abuse. 2022 Jan;23(1):288-300. doi: 10.1177/1524838020939126. Epub 2020 Jul 23. PMID 32700641
- [Background] Bratton, S., Ray, D., Rhine, T., & Jones, L. 2005. "The Efficacy of Play Therapy With Children: A Meta-Analytic Review of Treatment Outcomes," Professional Psychology: Research and Practice, 36, 376-390.
- [Background] Diaz-Rodriguez M, Alcantara-Rubio L, Aguilar-Garcia D, Perez-Munoz C, Carretero-Bravo J, Puertas-Cristobal E. The Effect of Play on Pain and Anxiety in Children in the Field of Nursing: A Systematic Review. J Pediatr Nurs. 2021 Nov-Dec;61:15-22. doi: 10.1016/j.pedn.2021.02.022. Epub 2021 Mar 10. PMID 33711642
- [Background] Nursanaa, W., Ady, I. 2020. "Play Therapy for Children with Anxiety Disorders," Proceedings of Social Sciences & Humanities, 81-86.
- [Background] Gülmez, İ., & Karaaziz, M. 2023. "A systematic review on the use of play therapy in sexually abused children," The Journal of Social Sciences, 62(62), 450-466.
- [Background] Leblanc, M., & Ritchie, M. 2001. "A meta-analysis of play therapy outcomes," Counselling Psychology Quarterly, 14, 149-163.
- [Background] Humble JJ, Summers NL, Villarreal V, Styck KM, Sullivan JR, Hechler JM, Warren BS. Child-Centered Play Therapy for Youths Who Have Experienced Trauma: a Systematic Literature Review. J Child Adolesc Trauma. 2018 Nov 9;12(3):365-375. doi: 10.1007/s40653-018-0235-7. eCollection 2019 Sep. PMID 32318206
- [Background] Ray, D. C., & Armstrong, S. A. 2021. "Child-centered play therapy: A review of research and practice," International Journal of Play Therapy, 30(1), 1-12.